CLINICAL TRIAL: NCT01565265
Title: Prospective Randomized Study Comparing Ovarian Stimulation With Pergoveris Supported by a GnRH Agonist in a Long Protocol Versus Multidose GnRH Antagonist Regimen in Young Infertile Women Treated With ICS
Brief Title: Comparing Ovarian Stimulation for Assisted Reproduction With Two Different Forms of Pituitary Suppression
Acronym: Pergoveris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBCH001; UBCH001 (Other Grant/Funding Number: University Hospital of Basel, Switzerland)
Record Dates: First submitted 2012-02-28; First posted 2012-03-28 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Female Infertility Due to Nonimplantation of Ovum; Complications Associated With Artificial Fertilization
Keywords: ovarian hyperstimulation; GnRH antagonist; GnRH agonist; assisted reproduction; FSH; LH
MeSH Terms: interventions — pergoveris; Gonadotropin-Releasing Hormone; cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GnRH agonist long protocol (Active Comparator): Pergoveris will be administered daily from cycle day 2 to ovulation induction together with decapeptyl, which will be administered from the midluteal phase of the preceding menstrual cycle up to ovulation induction.
  Interventions: Drug: Pergoveris in long protocol with GnRH agonist
- antagonist protocol (Experimental): Pergoveris will be administered daily from cycle day 2 to ovulation induction together with Cetrotide, which will be administered from the day six up to ovulation induction.
  Interventions: Drug: Pergoveris in GnRH antagonist protocol

INTERVENTIONS:
Drug: Pergoveris in long protocol with GnRH agonist — Ovarian hyperstimulation with recombinant FSH and recombinant FSH Ovulation induction with recombinant HCG Oocyte collection for ICSI
  Other Names: Pergoveris
  Arms: GnRH agonist long protocol
Drug: Pergoveris in GnRH antagonist protocol — Ovarian hyperstimulation with recombinant FSH and recombinant FSH Ovulation induction with recombinant HCG Oocyte collection for ICSI
  Other Names: Cetrotide
  Arms: antagonist protocol

SUMMARY:
The purpose of this study is to assess the non-inferiority of a multidose GnRH antagonist (cetrorelix) regimen to a GnRH agonist (triptorelin) long protocol in young infertile women undergoing ovarian stimulation with Pergoveris 150 I.U./75 I.U. (r-hFSH/ r-hLH) for ICSI treatment because of male infertility.

To assess the efficacy of ovarian stimulation using either a GnRH antagonist (cetrorelix) or a GnRH agonist (triptorelin) long protocol in infertile women with good prognosis and to determine the safety of ovarian stimulation.

Subsample analysis: in 10 patients of each of both arms, serum samples will be collected daily during the stimulation period and be stored frozen at -70 °C. The following hormone concentrations will be measured later in single assay batches: LH, FSH, oestradiol, progesterone, androstenedione, testosterone, inhibin A, inhibin B, AMH.

Multinational, multicentre, open label, randomized, 2-arm parallel-group phase IV study. Eligible patients will be randomly allocated to one of the two groups: the agonist group will receive Decapeptyl® 0.1 mg (triptorelin) starting in the mid-luteal phase of the natural cycle until downregulation until the day of ovulation induction. The antagonist group will receive cetrorelix 0.25 mg from stimulation day 6 to ovulation induction. In both groups, Pergoveris® 150 I.U./75 I.U. (r-hFSH/r-hLH) will be used for ovarian stimulation from cycle day 2 to ovulation induction.

DETAILED DESCRIPTION:
In assisted reproductive technology (ART), follicular growth is stimulated with exogenous gonadotropins to obtain multiple mature oocytes for fertilization. In a natural cycle, oocyte maturation and ovulation is triggered by endogenous luteinizing hormone (LH). To prevent a premature surge of LH and subsequent premature ovulation and cancellation of the ART cycle, a gonadotropin releasing hormone (GnRH) agonist is commonly used to inhibit endogenous gonadotropin release leading to premature ovulation or luteinization. After a short-term initial stimulation of the pituitary gland, continuous administration of a GnRH agonist leads to the downregulation of GnRH receptors of the pituitary and thus prevents synthesis and release of follicle-stimulating hormone (FSH) and LH from that organ.

Endogenous gonadotropin release may also be prevented by using GnRH antagonists instead of GnRH agonists. During the past decade, two GnRH antagonists (cetrorelix, ganirelix) have been licensed for prevention of premature LH surge and ovulation during ovarian hyperstimulation for assisted reproduction. The antagonist competes directly with the physiological GnRH for binding to the pituitary GnRH receptors and provides quicker suppression of gonadotropin release without the initial flare up. Compared with the GnRH agonist long protocol, GnRH antagonists require a considerably shorter treatment period, less exogenous gonadotropin for ovarian stimulation, and are associated with fewer side effects, and a lower risk of ovarian hyperstimulation syndrome (OHSS). An early meta-analysis from 2002, which included the first studies comparing GnRH agonist and antagonist treatment regimens, showed that clinical pregnancy was lower with GnRH antagonist treatment. However, there were no statistically significant differences in life-birth rate or in the probability of life birth between the protocols, as shown in a more recent review. However, GnRH agonists are still routinely used in most infertility centres, whereas GnRH antagonists are still preferentially prescribed to older women with unfavourable prognosis. The equivalence of both protocols has only been evaluated in ovarian hyperstimulation based on recombinant FSH only.

Another difference among both protocols consists of the sudden blockage of endogenous LH secretion caused by the administration of the GnRH antagonist, which is usually given when the follicles reach the size of 12 mm (around day 6 of the menstrual cycle). At that developmental stage, the LH receptor is present in the follicles participating in follicular function. In women treated with the long protocol, low endogenous levels of LH have been associated with low pregnancy rates. At present, conflicting data have been reported with regard to the effect of either low or high levels of LH during the midfollicular phase on the pregnancy rates, regardless whether GnRH agonists or GnRH antagonists were used. However, all these studies were performed with recombinant FSH lacking all LH activity and one single day measurement of LH concentration in the serum may not reflect the endocrine activity of LH throughout follicular development. The need for the presence of LH during follicular development has been demonstrated unequivocally in women suffering of hypogonadotropic ovarian failure (WHO I), which lead to the development of Pergoveris® 150 I.U./75 I.U.

Pergoveris® 150 I.U./75 I.U. is used to stimulate the development of follicles in the ovaries and was granted European marketing authorization in 2007. It consists of a fixed combination of recombinant human follicle-stimulating hormone (r-hFSH) and recombinant human luteinizing hormone (r-hLH) and allows the administration of both substances in a single injection. So far, no study has been performed to demonstrate the equivalence of Pergoveris® in the GnRH antagonist protocol as compared to the long protocol based on a GnRH agonist.

The current study aims to assess the non-inferiority of a multidose GnRH antagonist treatment regimen to a GnRH agonist long protocol in young infertile women (< 36 years) with good prognosis undergoing ovarian stimulation with Pergoveris® for intracytoplasmic sperm injection (ICSI) because of non-borderline male infertility. In addition, the safety of ovarian stimulation with Pergoveris will be evaluated for both treatment regimens, especially with regard to the incidence of OHSS.

The primary objective of this study is to assess the non-inferiority of a multidose GnRH antagonist (cetrorelix) regimen to a GnRH agonist (triptorelin) long protocol in young infertile women undergoing ovarian hyperstimulation with Pergoveris® 150 I.U./75 I.U. (r-hFSH/ r-hLH) for ICSI treatment because of male infertility. Non-inferiority is defined by the number of mature metaphase II oocytes available for ICSI.

Secondary objectives:

* To assess the efficacy of ovarian stimulation with Pergoveris using either a GnRH antagonist (cetrorelix) or a GnRH agonist (triptorelin) long protocol in infertile women with good prognosis with respect to the number of pregnancies achieved in each group.
* To determine the safety of ovarian stimulation with respect to the number of women suffering of the ovarian hyperstimulation syndrome (OHSS).

This is a clinical phase IV, multinational, multicentre study using an open label, randomized, 2-arm parallel-group design. The study will be conducted at various treatment units in Europe, including Switzerland (1 centre) and Israel.

Eligible patients will be randomly assigned to one of the two treatment arms:

* agonist group: r-hFSH/r-hLH 150 I.U./75 I.U. (Pergoveris®) daily from cycle day 2 to ovulation induction and triptorelin 0.1 mg daily from the mid-luteal phase (day 21 - 24) of the pre-ART cycle to ovulation induction.
* antagonist group: r-hFSH/r-hLH 150 I.U./75 I.U. (Pergoveris®) daily from cycle day 2 to ovulation induction and cetrorelix 0.25 mg daily from cycle day 7 (stimulation day 6) to ovulation induction.

ELIGIBILITY:
Inclusion Criteria:

Female patients younger than 36 years of age with an indication for ICSI:

* 20 to 35 years inclusive
* body mass index between 19 and 30 kg/m2
* indication for ICSI due to male infertility
* cycle length 27 to 32 days
* presence of both ovaries
* rubella immunity
* written informed consent

Exclusion Criteria:

* age > 35 years
* pregnancy and breast feeding
* ovarian endometriosis
* uterine fibroids interfering with endometrial proliferation
* sperm retrieval from the epididymis or the testis
* more than one previous ART treatment with pregnancy
* known or suspected hypersensitivity to active substances
* clinically relevant systemic disease
* previous enrollment to this study
* know or suspected non-compliance, drug or alcohol abuse

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
number of mature oocytes | up to two years
  The primary objective of this study is to assess the non-inferiority of a multidose GnRH antagonist (cetrorelix) regimen to a GnRH agonist (triptorelin) long protocol in young infertile women undergoing ovarian hyperstimulation with Pergoveris for ICSI treatment because of male infertility. Non-inferiority is defined by the number of mature metaphase II oocytes available for ICSI.

SECONDARY OUTCOMES:
incidence of ovarian hyperstimulation syndrome (OHSS) | up to two years
  The safety of ovarian stimulation with respect to the number of women suffering of the ovarian hyperstimulation syndrome (OHSS). OHSS is defined by enlargement of both ovaries together with ascites and haematocrit rise above 45%.
The number of early miscarriages. | up to two years
  Miscarriage is defined a pregnancy loss within 12 weeks after the last menstruation.
The number of participants with adverse events. | up to two years
  Adverse event is defined as any untoward medical occurrence in a patient or a clinical investigation subject, who was administerd a pharmaceutical product and which does not necessarily must have a causal relationship with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christian De Geter, Prof., Principal Investigator — University of Basel
Locations (1):
- University Hospital of Basel, Basel, Switzerland

REFERENCES:
- [Background] Kolibianakis EM, Collins J, Tarlatzis BC, Devroey P, Diedrich K, Griesinger G. Among patients treated for IVF with gonadotrophins and GnRH analogues, is the probability of live birth dependent on the type of analogue used? A systematic review and meta-analysis. Hum Reprod Update. 2006 Nov-Dec;12(6):651-71. doi: 10.1093/humupd/dml038. Epub 2006 Aug 18. PMID 16920869
- [Background] Kolibianakis EM, Zikopoulos K, Schiettecatte J, Smitz J, Tournaye H, Camus M, Van Steirteghem AC, Devroey P. Profound LH suppression after GnRH antagonist administration is associated with a significantly higher ongoing pregnancy rate in IVF. Hum Reprod. 2004 Nov;19(11):2490-6. doi: 10.1093/humrep/deh471. Epub 2004 Aug 19. PMID 15319383
- [Background] Al-Inany H, Aboulghar M. GnRH antagonist in assisted reproduction: a Cochrane review. Hum Reprod. 2002 Apr;17(4):874-85. doi: 10.1093/humrep/17.4.874. PMID 11925376
- [Background] Pouly JL, Bachelot A, de Mouzon J, Devaux A; FIVNAT. [Comparison of agonists versus antagonists for i.v.f. stimulation: the French FIVNAT survey 2001-2002]. Gynecol Obstet Fertil. 2004 Sep;32(9):737-40. doi: 10.1016/j.gyobfe.2004.07.011. French. PMID 15380755
- [Background] Griesinger G, Felberbaum R, Diedrich K. GnRH antagonists in ovarian stimulation: a treatment regimen of clinicians' second choice? Data from the German national IVF registry. Hum Reprod. 2005 Sep;20(9):2373-5. doi: 10.1093/humrep/dei086. Epub 2005 Jun 2. PMID 15932915
- [Background] Huirne JA, Hugues JN, Pirard C, Fischl F, Sage JC, Pouly JL, Obruca A, Braat DM, van Loenen AC, Lambalk CB. Cetrorelix in an oral contraceptive-pretreated stimulation cycle compared with buserelin in IVF/ICSI patients treated with r-hFSH: a randomized, multicentre, phase IIIb study. Hum Reprod. 2006 Jun;21(6):1408-15. doi: 10.1093/humrep/del030. Epub 2006 Mar 14. PMID 16537563
- [Background] Penarrubia J, Fabregues F, Creus M, Manau D, Casamitjana R, Guimera M, Carmona F, Vanrell JA, Balasch J. LH serum levels during ovarian stimulation as predictors of ovarian response and assisted reproduction outcome in down-regulated women stimulated with recombinant FSH. Hum Reprod. 2003 Dec;18(12):2689-97. doi: 10.1093/humrep/deg506. PMID 14645193
- [Background] Coppola F, Poti ER, Barusi L, Ferrari B, Salvarani MC, Vadora E. Profound luteinizing hormone suppression induces a deleterious follicular environment during assisted reproduction technology. Fertil Steril. 2003 Feb;79(2):459-60. doi: 10.1016/s0015-0282(02)04671-x. No abstract available. PMID 12568871
- [Background] Merviel P, Antoine JM, Mathieu E, Millot F, Mandelbaum J, Uzan S. Luteinizing hormone concentrations after gonadotropin-releasing hormone antagonist administration do not influence pregnancy rates in in vitro fertilization-embryo transfer. Fertil Steril. 2004 Jul;82(1):119-25. doi: 10.1016/j.fertnstert.2003.11.040. PMID 15236999
- [Background] Burgues S; Spanish Collaborative Group on Female Hypogonadotrophic Hypogonadism. The effectiveness and safety of recombinant human LH to support follicular development induced by recombinant human FSH in WHO group I anovulation: evidence from a multicentre study in Spain. Hum Reprod. 2001 Dec;16(12):2525-32. doi: 10.1093/humrep/16.12.2525. PMID 11726569
- [Background] Recombinant human luteinizing hormone (LH) to support recombinant human follicle-stimulating hormone (FSH)-induced follicular development in LH- and FSH-deficient anovulatory women: a dose-finding study. The European Recombinant Human LH Study Group. J Clin Endocrinol Metab. 1998 May;83(5):1507-14. doi: 10.1210/jcem.83.5.4770. PMID 9589647